CLINICAL TRIAL: NCT01584115
Title: Phase I Clinical Trial of a Therapeutic Vaccine for Malignancies, Comprising the Tumor Antigen NY-ESO-1 in Combination With the Adjuvant MPLA of Bordetella Pertussis. Evaluation of Toxicity and Immunogenicity
Brief Title: Clinical Trial of a Therapeutic Vaccine With NY-ESO-1 in Combination With the Adjuvant Monophosphoryl Lipid A (MPLA)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Instituto de Investigação em Imunologia (Other)
Collaborators: Butantan Institute (Other Government)
Responsible Party: Principal Investigator, Pedro Giavina-Bianchi, Principal Investigator, Instituto de Investigação em Imunologia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6889; CNPq 577582/2008-9 (Other Grant/Funding Number: CNPq 577582/2008-9)
Record Dates: First submitted 2012-04-21; First posted 2012-04-24 (Estimated); Last update posted 2012-04-25 (Estimated); Status verified 2012-04

CONDITIONS: Cancer.; Melanoma.; Ovarian Cancer.; Lung Cancer.
Keywords: Cancer.; Melanoma.; Ovarian cancer.; Lung cancer.; NY-ESO-1.; MPLA (monophosphoryl lipid A).; Tumor antigen.; Bordetella pertussis.
MeSH Terms: conditions — Neoplasms; Melanoma; Ovarian Neoplasms; Lung Neoplasms | interventions — monophosphoryl lipid A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- NY-ESO-1 (Experimental): NY-ESO-1 combined with MPLA vaccine
  Interventions: Biological: NY-ESO-1 combined with MPLA; Biological: NY-ESO-1 combined with MPLA vaccine

INTERVENTIONS:
Biological: NY-ESO-1 combined with MPLA — Each patient will receive six doses of the formulation, administered intra-muscular, with an interval of 4 weeks between doses, and the first immunization performed 6 weeks after the completion of standard treatment. NY-ESO-1 (250 mcg) amd MPLA (100 mcg).
Biological: NY-ESO-1 combined with MPLA vaccine — Immunization os cancer patients with NY-ESO-1 combined with MPLA vaccine

SUMMARY:
This study is a clinical trial phase I/II. Its goal is to determine the safety, tolerability, immunogenicity and efficacy of a therapeutic vaccine with the tumor antigen NY-ESO-1 combined with the adjuvant MPLA from B. pertussis in cancer patients.

DETAILED DESCRIPTION:
The safety and immunogenicity of the vaccine with the antigen NY-ESO-1 in combination with the MPLA will be evaluated in a phase 1 clinical trial conducted in patients with malignancies that express the antigen (lung, ovarian and melanoma). This study will involve 15 patients, who will receive 250 mcg of NY-ESO-1 and 100 mcg of MPLA.

ELIGIBILITY:
Inclusion Criteria:

* In this study, will be included fifteen patients aged over 18 years, with a confirmed diagnosis of malignant neoplasms, which have proven NY-ESO-1 expression by immunohistochemistry and have undergone the standard treatment.

Exclusion Criteria:

* Will be excluded from the study patients with continuous use of systemic steroids, immunosuppressive agents and antibiotics, and with severe chronic systemic disease.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2012-07; Primary Completion 2013-07 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Safety | Six months after immunization.
  CTCAE (Common Terminology Criteria for Adverse Events)

SECONDARY OUTCOMES:
Immunogenicity | Six months after immunization.
  IgG against NY-ESO-1 (ELISA). NY-ESO-1-specific T cells CD4+ and CD8+ (ELISPOT and FACs - flow citometry with tetramers).

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Giavina-Bianchi, MD,PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- Hospital das Clinicas da FMUSP, São Paulo, Brazil